CLINICAL TRIAL: NCT02557230
Title: Malignant Genito-urinary Tumors in Children: South Egypt Cancer Institute Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Ped GU Tumors
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Genitourinary Neoplasms; Neoplasms, Genitourinary
Keywords: Childhood Cancer; Genitourinary tumors; urogenital tumors; Pediatric Oncology
MeSH Terms: conditions — Urogenital Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify demographic & disease characteristics in pediatric oncology patients diagnosed with one of genitourinary tumors & treatment outcomes in these patients.

DETAILED DESCRIPTION:
Background:

Tumors of the kidney, bladder, prostate, testis, and adrenal represent a large part of the adult urologic practice, but are relatively infrequent in children.

Genitourinary tumors contribute to pediatric solid tumors. Wilms tumor, rhabdomyosarcoma, and germ cell tumors are the most common malignant genitourinary tumors in children.

The natural history and management of these tumors in the pediatric age is different from that of the adults. As result of the successful work of several clinical trial groups in recent decades, there has been a significant improvement in their cure rates.

Patients & Methods:

From January 2001 till December 2015, retrieval & analysis of the medical records of pediatric patients with genitourinary tumors will be made at the pediatric oncology department, South Egypt Cancer Institute which represents the largest referral center in Upper Egypt. These data will be categorized according to demographic characteristics, clinico-pathologic features, treatment modalities received, and outcomes of treatments in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than or equal to 18 years.
* Patients diagnosed with any of neoplasms affecting the genitourinary system.

Exclusion Criteria:

* Patients whose age more than 18 years.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with any of genitourinary neoplasms, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Denes FT, Duarte RJ, Cristofani LM, Lopes RI. Pediatric genitourinary oncology. Front Pediatr. 2013 Dec 16;1:48. doi: 10.3389/fped.2013.00048. PMID 24400293
- [Background] Lambert S. Adult Survivors of Pediatric Genitourinary Tumors. In: Wood HM, Wood D, editors. Transition and Lifelong Care in Congenital Urology: Springer International Publishing; 2015. p. 209-16.